CLINICAL TRIAL: NCT05472194
Title: Promoting Inclusive Education Through Executive Functions - Study Protocol of a Randomized Control Trial
Brief Title: Promoting Inclusive Education Through Executive Functions
Acronym: EduFun
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Sonia Sousa, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EduFun2022
Record Dates: First submitted 2022-06-23; First posted 2022-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Training
Keywords: Inclusive Education; Executive Functions; Cognitive Tools

STUDY DESIGN:
Intervention Model Description: The protocol includes a randomized controlled trial with a follow-up at six months involving two groups per age range (5,6 and 7Y) -a training group, which will be enrolled in the InSchool program and an active control group that will be participating in the regular kindergarten/elementary school activities. Participants will be randomly assigned to each group to control for inter-individual variability in executive functions' developmental level, which could distinctly impact the study results.
Who Masked: Participant
Masking Description: Participants will be randomly assigned for the experimental or control group with no information on the nature of the group they will be assigned. Additionally, no information about the training activities will be passed on to the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Experimental): Participants allocated to the Experimental condition will be following a cognitive training program using a set of game-based activities specifically developed to train executive functions.
  Interventions: Behavioral: InSchool Training Program
- Control Condition (Active Comparator): Participants allocated to the Control condition will be following the same sessions of the training program (similar to the Experimental group) while playing with a set of commonly used games within the school context (e.g. puzzles).
  Interventions: Behavioral: Regular school activities

INTERVENTIONS:
Behavioral: InSchool Training Program — The goal of the intervention is to promote and boost the development of executive functions in preschool and elementary school-aged children by means of engagement in meaningful and challenging activities. The method to achieve this consists on weekly intervention sessions run by teachers with a set of games specially developed to train executive functions.
  Arms: Experimental Condition
Behavioral: Regular school activities — Children in the control group will be playing with the regular school activities.
  Arms: Control Condition

SUMMARY:
Background: Recently governments worldwide have been doing enormous efforts to ensuring egalitarian educational opportunities for all children. However, the number of children that remain out of the school or lack proficiency in academic performance is still very worrying. One of the factors that seems to contribute to such inequalities is socioeconomic status (SES). SES strongly impacts the developmental trajectory of both the brain and cognitive abilities as off early childhood, further affecting learning and academic success.

Despite the great interest in building inclusive societies and the promising results of executive functions' training programs for leveling the SES-achievement disparities, only a few studies have actually included schools from low-SES settings and lack a comprehensive, evidence-based background underlying the intervention protocols. Thus, with a preventive emphasis, the current project aims to implementing and evaluating a cost-effective game-based training protocol to promote and boost the development of executive functions in preschool and elementary school-aged children from disadvantaged contexts, ultimately contributing to prevent school dropout and reduce academic inequalities.

DETAILED DESCRIPTION:
A randomized controlled trial will be implemented in Portuguese schools embedded in low-income settings. It will include a total of 396 participants, 132 per age group: 5,6 and 7 years old. At each age group a total of 132 children will be enrolled in the program for 4 weeks, 66 in the active control group, and 66 in the intervention group. The assessment protocol will include demographics, including SES, and evaluation of executive functions. Both groups -control and intervention- will complete the same assessment protocol at three distinct moments -baseline, post-intervention, and 6 months' follow-up. The training program will comprise the following: (i) 3 weekly sessions of 30 minutes each (ii) each session will be dedicated to train a specific domain of executive functions -working memory, inhibition and cognitive flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Typically developed children of 5, 6, and 7 years old attending the regular curriculum at public educational services -kindergarten and elementary school.

Exclusion Criteria:

* Presence or history of cognitive deficits, neurological or psychiatric condition.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12-09 (Estimated); Study Completion 2027-12-09 (Estimated)

PRIMARY OUTCOMES:
Executive functions (Working memory) | Through study completion, an average of 1 year.
  Accuracy, measured through the number of hits, will be collected from the participant's performance on a working memory task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.
Executive functions (Working memory) | Through study completion, an average of 1 year.
  Reaction times, measured as seconds needed to give a response, will be collected from the participant's performance on a working memory task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.
Executive functions (Inhibitory control) | Through study completion, an average of 1 year.
  Accuracy, measured through the number of hits, will be collected from the participant's performance on an inhibitory control task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.
Executive functions (Inhibitory control) | Through study completion, an average of 1 year.
  Reaction times, measured as seconds needed to give a response, will be collected from the participant's performance on an inhibitory control task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.
Executive functions (set shifting) | Through study completion, an average of 1 year.
  Accuracy, measured through the number of hits, will be collected from the participant's performance on a set shifting task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.
Executive functions (set shifting) | Through study completion, an average of 1 year.
  Reaction times, measured as seconds needed to give a response, will be collected from the participant's performance on a set shifting task, conducted using a digital platform specifically built to assess the hypothetical differences in participant's level of achievement between the pretest and posttest assessments.

SECONDARY OUTCOMES:
School Grades | Through study completion, an average of 1 year.
  Grades in math and Portuguese of each participant's current school year are the secondary outcomes and will be requested to their teachers. This measure will be applicable only to the 6 and 7 years old children.

CONTACTS AND LOCATIONS:
Overall Officials: Sónia Sousa, PhD, Principal Investigator — School of Psychology, University of Minho